CLINICAL TRIAL: NCT03927820
Title: A Pharmacist-Led Intervention to Increase Inhaler Access and Reduce Hospital Readmissions (PILLAR)
Acronym: PILLAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Tate Davis, Clinical Pharmacist, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PILLAR
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: COPD; Asthma
Keywords: inhaler; pharmacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist Intervention (Active Comparator): Patients randomized to the intervention arm received usual care plus inhaler review by study pharmacist who made recommendations for inhaler changes based on clinical guideline and insurance formulary compliance. Recommendations were sent to the patient's team for final approval prior to discharge.
  Interventions: Other: Benefits investigation
- Usual Care (No Intervention): Patients randomized to the usual care arm received care by the primary team which includes an inpatient pharmacist who does not have access to benefits investigation technology. The study pharmacist was not involved to review inhalers for optimization prior to discharge.

INTERVENTIONS:
Other: Benefits investigation — The study pharmacist will review the prescribed inhaler for 1) insurance coverage and 2) clinical appropriateness. The pharmacist will conduct a benefits investigation at time of hospital admission. The benefits investigation involves running test claims for inhalers to determine the most cost-effective inhaler for the patient's insurance plan. The study pharmacist will utilize clinical practice guidelines to assess appropriateness of the prescribed inhaler. Based on this review, the study pharmacist will submit a pharmacy consult to the inpatient pharmacist on the patient's healthcare team who will pend the inhaler orders (changing the patient's prescribed inhaler, if necessary) for the prescriber to send to the Meds to Beds discharge pharmacy. The Meds to Beds pharmacist will counsel the patient on inhaler use techniques prior to discharge.
  Arms: Pharmacist Intervention

SUMMARY:
The goal of this study is to assess the impact of pharmacist-led benefits investigations and application of clinical practice guidelines on patient access to inhalers and time to hospital readmission or Emergency Department (ED) visit.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient admitted to Vanderbilt University Medical Center (VUMC) (excluding surgery services)
* on a long acting inhaler or prescribed a long acting inhaler during admission.

Exclusion Criteria:

* Diagnosis of cystic fibrosis
* Diagnosis of graft versus host disease (GVHD)
* no medication insurance
* discharge to any post-acute care facility or inpatient hospice
* death during hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 914 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time to either hospital readmission or ER visit | 6 months
  Combined time (days) to either hospital readmission or emergency department visit after hospitalization (all outcomes measured at 6 months post-discharge with a 3 month interim analysis)

SECONDARY OUTCOMES:
Frequency of ED visit | 6 months
  number of ED visits 6 months post-discharge
frequency of hospital readmissions | 6 months
  number of hospital readmission 6 months post-discharge
time to 1st ED visit (days) | 6 months
  time until the first ED visit post-discharge
time to 1st readmission (days) | 6 months
  time until the first readmission post-discharge
frequency of prescribed inhaler at discharge | 6 months
  number of times the recommended inhaler was prescribed at discharge
frequency of short course prescription of oral steroid | 6 months
  number of oral steroid prescriptions in the 6 months post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Niehoff, PharmD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Univeristy Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No